CLINICAL TRIAL: NCT00871650
Title: Neurobiological Correlates of PTSD During REM Sleep (REM-P)
Brief Title: Neurobiological Correlates of Post Traumatic Stress Disorder (PTSD) During Rapid Eye Movement (REM) Sleep
Acronym: REM-P
Status: Completed | Type: Observational
Sponsor: University of Pittsburgh (Other)
Responsible Party: Sponsor
Other Study IDs: MH083035-01
Record Dates: First submitted 2009-03-26; First posted 2009-03-30 (Estimated); Last update posted 2013-01-16 (Estimated); Status verified 2013-01

CONDITIONS: Post-Traumatic Stress Disorder
Keywords: Post Traumatic Stress Disorder; PTSD; Brain; Imaging; PET; Neural; Sleep; REM Sleep
MeSH Terms: conditions — Stress Disorders, Post-Traumatic

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Combat Veterans with PTSD: Male Veterans of Operation Iraqi Freedom (OIF) and/or Operation Enduring Freedom (OEF), ages 18-50, with Combat Exposure Scale score > 17, who are not on medication and do not have trauma history before age 18.
  Interventions: Other: Sleep data recording; Other: PET scan - waking; Other: PET scan - REM Sleep
- Combat Veterans without PTSD: Male Veterans of Operation Iraqi Freedom (OIF) and/or Operation Enduring Freedom (OEF), ages 18-50, with combat experience, who are not suffering from PTSD, and who are not on medication.
  Interventions: Other: Sleep data recording; Other: PET scan - waking; Other: PET scan - REM Sleep

INTERVENTIONS:
Other: Sleep data recording — After completing the screening procedures, eligible participants will sleep in the laboratory for three consecutive nights of EEG sleep studies, one waking [18F]-FDG PET scan, and one REM sleep PET scan according to published methods.
Other: PET scan - waking — After completing the screening procedures, eligible participants will sleep in the laboratory for three consecutive nights of EEG sleep studies, one waking [18F]-FDG PET scan, and one REM sleep PET scan according to published methods.
Other: PET scan - REM Sleep — After completing the screening procedures, eligible participants will sleep in the laboratory for three consecutive nights of EEG sleep studies, one waking [18F]-FDG PET scan, and one REM sleep PET scan according to published methods.

SUMMARY:
The overarching aim of this Exploratory/Developmental Research Grant Award (R21) is to explore the neurobiological correlates of PTSD during REM sleep by using state-of-the science positron emission tomography (PET) sleep imaging. This study will allow us to gain insight into the differences in sleep and waking brain mechanisms between veterans with PTSD and those without PTSD.

ELIGIBILITY:
General Inclusion Criteria:

* Male OIF/OEF returnees between the ages of 18 and 45 years old
* Combat Exposure Scale score > 17
* Not taking medications known to affect sleep or wake function for at least 2 weeks (6 weeks for fluoxetine).
* No history of trauma before age 18

Specific Inclusion Criteria for Subjects with PTSD:

* Meet diagnostic criteria for current PTSD according to the CAPS-1
* CAPS-1 score is less than 80

Specific Inclusion Criteria for Subjects without PTSD:

* Total CAPS-1 scores < 17
* Does not meet criteria for PTSD

Exclusion Criteria:

* Trauma occurred less than 3 months prior to study entry
* CES score < 17
* Taking medications known to affect sleep and / or brain glucose metabolism
* Current diagnosis of depression as determined by the SCID or BDI score > 13
* History of psychotic or bipolar disorder
* Current history (within 3 months) of substance or alcohol abuse as determined by the SCID
* Positive alcohol blood test at screening or during the PET protocol
* Significant or unstable acute or chronic medical conditions
* Other current sleep disorders, such as insufficient sleep syndrome, delayed sleep phase syndrome, narcolepsy, restless legs syndrome, periodic leg movement disorder, obstructive sleep apnea, and current night shift work, suspected during the structured interview. Individuals who are found to have a apnea-hypopnea index (AHI) > 10 or an index of periodic leg movements with arousal > 15 will be excluded.
* Presence of implanted devices such as cardiac pacemaker, aneurysm clip, ear implant, shrapnel, neurostimulators or other metal devices
* Fear of closed spaces
* Previous radiation. Due to the risk of radiation exposure, we will exclude subjects who have had PET scans or other radiotracer exposure in the previous year.
* History of open head injury.

Ages: 18 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Male Veterans of Operation Iraqi Freedom (OIF) and/or Operation Enduring Freedom (OEF), ages 18-50, with combat experience, who are not on medication.
Sampling Method: Non-Probability Sample
Enrollment: 24 (Estimated)
Dates: Start 2009-03; Primary Completion 2011-03 (Actual); Study Completion 2011-11 (Actual)

PRIMARY OUTCOMES:
Brain glucose metabolism | During waking
Brain glucose metabolism | During REM sleep

CONTACTS AND LOCATIONS:
Locations (1):
- University of Pittsburgh, Pittsburgh, Pennsylvania, United States

REFERENCES:
- [Derived] Stocker RP, Cieply MA, Paul B, Khan H, Henry L, Kontos AP, Germain A. Combat-related blast exposure and traumatic brain injury influence brain glucose metabolism during REM sleep in military veterans. Neuroimage. 2014 Oct 1;99:207-14. doi: 10.1016/j.neuroimage.2014.05.067. Epub 2014 Jun 2. PMID 24893322